CLINICAL TRIAL: NCT07108673
Title: Value of Voxel-Based Morphometry in Assessing Brain Structural Abnormalities in Schizophrenia and Nicotine Use Disorder.
Brief Title: Value of Voxel-Based Morphometry in Schizophrenia
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hesham Mohammed Abdel-Moty, Prinicipal investigator, Assiut University
Other Study IDs: NCTMRISCHIZ2025
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia
Keywords: Voxel-Based Morphometry; Brain Structural Abnormalities; Schizophrenia; Nicotine use disorder
MeSH Terms: conditions — Schizophrenia; Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Schizophrenic patients without nicotine dependence
  Interventions: Diagnostic Test: MRI
- Schizophrenic patients with nicotine dependence
  Interventions: Diagnostic Test: MRI
- Individuals with nicotine dependence but without schizophrenia
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — structural MRI imaging and behavioral testing (e.g. Barratt Impulsiveness scale) both performed by skilled physicians.

SUMMARY:
This cross-sectional observational study investigates structural brain abnormalities in schizophrenia and nicotine use disorder (NUD), with a focus on understanding how these abnormalities correlate with behavioral traits such as decision-making and impulsivity. Schizophrenia is often associated with reduced gray matter (GM) in the prefrontal cortex and anterior cingulate cortex, while nicotine dependence is linked to changes in brain regions involved in reward processing. Nicotine use is particularly prevalent among individuals with schizophrenia, potentially compounding cognitive impairments.

Voxel-Based Morphometry (VBM), an advanced neuroimaging analysis technique, allows for the detection of subtle structural changes in the brain using MRI data. This study aims to utilize VBM to explore GM alterations in three participant groups:

Schizophrenic patients without nicotine dependence

Schizophrenic patients with nicotine dependence

Individuals with nicotine dependence but without schizophrenia

Each group will include 32 participants, making a total sample of 96, calculated using G*Power software assuming a medium effect size, alpha 0.05, and power 0.8. Inclusion criteria include confirmed diagnoses based on DSM-5 and the Fagerström Test for Nicotine Dependence, age 18-60, and MRI compatibility. Exclusion criteria involve other psychiatric or neurological disorders, substance use other than nicotine, and MRI contraindications.

Participants will undergo:

Structural MRI scans

Behavioral assessment using the Barratt Impulsiveness Scale

Clinical interviews using the Structured Clinical Interview for DSM-5

The primary outcome is to identify distinct patterns of GM reduction or alteration across groups, especially in regions involved in decision-making (e.g., prefrontal cortex, anterior cingulate cortex) and reward processing (e.g., ventral striatum). Secondary outcomes include correlating these structural findings with impulsivity and decision-making patterns.

Statistical analysis will be performed using SPSS v26. ANOVA will be used for quantitative comparisons across the three groups, while Chi-square or Fisher's exact tests will compare categorical variables. Pearson's correlation will be used to explore associations between brain changes and behavioral traits. A p-value <0.05 will be considered significant.

DETAILED DESCRIPTION:
Schizophrenia and nicotine use disorder are two conditions linked in part to distinct brain structural abnormalities that can significantly impact cognitive and behavioral functions, particularly in areas like decision-making and impulsivity. Schizophrenia (although it's exact cause is unknown) is often associated with reduced gray matter (GM) in regions such as the prefrontal cortex and anterior cingulate cortex, which are crucial for cognitive control and decision-making processes . Nicotine use disorder, on the other hand, has been linked to structural changes in brain areas involved in reward processing and impulsivity regulation. The overlap of these conditions is notable, as nicotine addiction is highly prevalent among schizophrenic patients, potentially exacerbating cognitive and behavioral dysfunctions .

Voxel-Based Morphometry (VBM) is a widely used neuroimaging technique that enables researchers to detect and quantify brain structural differences, particularly in GM, by analyzing MRI scans. VBM allows for the identification of subtle brain abnormalities that may contribute to the development of schizophrenia and nicotine dependence. These structural changes may provide insight into associated behavioral traits such as impaired decision-making and increased impulsivity, both of which are commonly observed in individuals with either or both conditions

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed schizophrenia (for groups 1 and 2).
* Nicotine dependence as defined by the Fagerström Test for Nicotine Dependence (for groups 2 and 3).
* Age range: 18-60 years.
* Schizophrenic patients must be stable on medications for at least 2 months.
* Written informed consent (from the patient or his carer).

Exclusion Criteria:

* History of other neurological or other psychiatric disorders (besides schizophrenia or nicotine dependence).
* Current substance use disorders other than nicotine.
* Severe head trauma or other conditions likely to affect brain structure.
* IQ below 70.
* MRI contraindications such as metallic implants (e.g. pace maker), claustrophobia or anxiety disorders severe enough to prevent comfortable MRI scanning will also be exclusion criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The targeted study groups are:
  Group 1: Schizophrenic patients without nicotine dependence. Group 2: Schizophrenic patients with nicotine dependence. Group 3: Nicotine use disorder individuals without schizophrenia.
  Each group will be matched for age, gender, and educational background to minimize potential confounding variables.
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
structural abnormalities by MRI | at the enrollment
  we will catch any structural abnormalities like GM reductions in the prefrontal cortex and anterior cingulate cortex

SECONDARY OUTCOMES:
Behavioral testing | at the enrollment
  Behavioral testing is expected to reveal that GM abnormalities correlate with impaired decision-making and increased impulsivity. By using Fagerstrom Test for Nicotine Dependence (FTND): Classifies participants' nicotine addiction levels.
  Structured Clinical Interview for DSM-5: Confirms diagnoses of schizophrenia and nicotine use disorder.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Du X, Choa FS, Chiappelli J, Bruce H, Kvarta M, Summerfelt A, Ma Y, Regenold WT, Walton K, Wittenberg GF, Hare S, Gao S, van der Vaart A, Zhao Z, Chen S, Kochunov P, Hong LE. Combining neuroimaging and brain stimulation to test alternative causal pathways for nicotine addiction in schizophrenia. Brain Stimul. 2024 Mar-Apr;17(2):324-332. doi: 10.1016/j.brs.2024.02.020. Epub 2024 Mar 5. PMID 38453003
- [Background] Wilke M, Kaufmann C, Grabner A, Putz B, Wetter TC, Auer DP. Gray matter-changes and correlates of disease severity in schizophrenia: a statistical parametric mapping study. Neuroimage. 2001 May;13(5):814-24. doi: 10.1006/nimg.2001.0751. PMID 11304078
- [Background] Liu H, Guan L, Nie Y, Li Q, Xue J, Yang Y, Rong S, Liang J, Guan Y, Zhai F, Ren Y, An Z, Dong Z, Han Z. Brain Magnetic Resonance Imaging Features of Nicotine-Dependent Individuals and Its Correlation with Polymorphisms of Dopamine D Receptor Gene. Contrast Media Mol Imaging. 2022 Aug 24;2022:2296776. doi: 10.1155/2022/2296776. eCollection 2022. PMID 36082055
- [Background] Brown GG, Lee JS, Strigo IA, Caligiuri MP, Meloy MJ, Lohr J. Voxel-based morphometry of patients with schizophrenia or bipolar I disorder: a matched control study. Psychiatry Res. 2011 Nov 30;194(2):149-56. doi: 10.1016/j.pscychresns.2011.05.005. Epub 2011 Sep 15. PMID 21924872
- [Background] Segall JM, Turner JA, van Erp TG, White T, Bockholt HJ, Gollub RL, Ho BC, Magnotta V, Jung RE, McCarley RW, Schulz SC, Lauriello J, Clark VP, Voyvodic JT, Diaz MT, Calhoun VD. Voxel-based morphometric multisite collaborative study on schizophrenia. Schizophr Bull. 2009 Jan;35(1):82-95. doi: 10.1093/schbul/sbn150. Epub 2008 Nov 7. PMID 18997157